CLINICAL TRIAL: NCT00627653
Title: PET (Positron Emission Tomography) Detection of the Effects of Aging on the Human Heart (Aim #2 Effect of a PPAR-Alpha Agonist on the Age Related Changes in Myocardial Metabolism and Mechanical Function)
Brief Title: Effect of a PPAR-Alpha Agonist on the Age Related Changes in Myocardial Metabolism and Mechanical Function
Acronym: PPAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Robert Gropler, MD, Washington University in St Louis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG0093; ROI AG15466
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Diseases
Keywords: PPAR; PET study; heart metabolism
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: fenofibrate — 148mg daily for 30 days
  Other Names: Lofibra; TriCor

SUMMARY:
The purpose of this study is to determine if treatment with a drug called fenofibrate, which is a PPAR-alpha agonist and controls how the heart metabolizes fats, will reverse the age-related decline in cardiac fat metabolism and mechanical function.

DETAILED DESCRIPTION:
In older Americans, cardiovascular disease is the leading cause of death and disability. It has been shown recently that with aging the human heart exhibits a decline in myocardial fatty acid utilization (MFAU) and oxidation (MFAO) and that these metabolic changes are paralleled by a decline in mechanical function. It has also been shown that peroxisome proliferator activated receptor alpha (PPAR-alpha) activates the expression of the genes encoding enzymes involved in mitochondrial fatty acid transport and oxidation. There is both indirect and direct evidence that PPAR-alpha-mediated responses decrease with age. Consequently, we hypothesize that changes in fatty acid in the aging heart may be mediated, at least in part, via a decline in PPAR-alpha-mediated responses. Thus, administration of a PPAR-alpha agonist to older humans will result in a shift in cardiac fatty acid metabolism to that more closely seen in younger humans and this shift will be paralleled by an improvement in cardiac mechanical function.

To prove or disprove this hypothesis, we will determine, in aged and young healthy volunteers, whether stimulation of PPAR-alpha using the partial agonist, fenofibrate, shifts myocardial substrate utilization by increasing MFAU and MFAO, and whether these changes are associated with an increase in left ventricular function. Study participants will have 4 clinic visits, each lasting approximately 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-75 or 21-35
* Normal glucose tolerance test
* Normal plasma fasting lipid panel (fasting total cholesterol less than 220 mg/dL)
* Normal rest/stress echocardiogram
* BMI (body mass index) less than 30 kg/m2
* Must be sedentary (active, but do not engage in regular exercise or jobs that require strenuous exertion)

Exclusion Criteria:

* Coronary artery disease
* High blood pressure
* Current smoker
* Diabetes mellitus
* Cardiovascular disease (signs and symptoms of any kind)
* Pregnant or breastfeeding

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Shift in Myocardial substrate utilization in aging hearts | After the day-30 PET scan

SECONDARY OUTCOMES:
Increased left ventricular function due to shift in substrate use in aging hearts | After the day-30 PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gropler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Ogawa T, Spina RJ, Martin WH 3rd, Kohrt WM, Schechtman KB, Holloszy JO, Ehsani AA. Effects of aging, sex, and physical training on cardiovascular responses to exercise. Circulation. 1992 Aug;86(2):494-503. doi: 10.1161/01.cir.86.2.494. PMID 1638717
- [Background] Coughlin SS, Neaton JD, Sengupta A, Kuller LH. Predictors of mortality from idiopathic dilated cardiomyopathy in 356,222 men screened for the Multiple Risk Factor Intervention Trial. Am J Epidemiol. 1994 Jan 15;139(2):166-72. doi: 10.1093/oxfordjournals.aje.a116978. PMID 8296783
- [Background] Haldeman GA, Croft JB, Giles WH, Rashidee A. Hospitalization of patients with heart failure: National Hospital Discharge Survey, 1985 to 1995. Am Heart J. 1999 Feb;137(2):352-60. doi: 10.1053/hj.1999.v137.95495. PMID 9924171
- [Background] Olivetti G, Melissari M, Capasso JM, Anversa P. Cardiomyopathy of the aging human heart. Myocyte loss and reactive cellular hypertrophy. Circ Res. 1991 Jun;68(6):1560-8. doi: 10.1161/01.res.68.6.1560. PMID 2036710
- [Background] Kannel WB, Belanger AJ. Epidemiology of heart failure. Am Heart J. 1991 Mar;121(3 Pt 1):951-7. doi: 10.1016/0002-8703(91)90225-7. PMID 2000773